CLINICAL TRIAL: NCT05642949
Title: Phase 1/2, Multi-center, Open-label, Dose Escalation and Cohort Expansion Study to Evaluate the Safety/Tolerability, Pharmacokinetics and Efficacy of MHB036C in Participants With Advanced or Metastatic Solid Tumors
Brief Title: Study of MHB036C in Participants With Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MHB036C-CP001EN
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Single group, but in two study parts, therefore two sequential arms are identified
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation - All Participants (Experimental): All participants enrolled in the dose escalation part.
  Interventions: Drug: MHB036C
- Dose Expansion - All Participants (Experimental): All participants enrolled in the dose expansion part
  Interventions: Drug: MHB036C

INTERVENTIONS:
Drug: MHB036C — MHB036C will be administered intravenously at a frequency of once every 3 weeks (Q3W).

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and anti-tumor efficacy of MHB036C in participants with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study is the first-in-human (FIH) trial of MHB036C, and contains two parts: dose escalation phase (part one) and dose expansion phase (part two).

The dose escalation phase is an open-label, multi-center study in which eligible participants with advanced or metastatic solid tumors will be enrolled to receive MHB036C monotherapy. This study is designed to assess the safety and tolerability of MHB036C in participants with advanced or metastatic solid tumors, to determine the maximum tolerated dose (MTD) of MHB036C, and to assess its pharmacokinetic profile and preliminary efficacy.

The dose expansion part is an open-label, multi-center, multi-cohort expansion study in which participants with advanced or metastatic solid tumors of some predefined cancer types will be enrolled to receive MHB036C monotherapy. Participants with same types of solid tumors will be randomized assigned into different selected dose groups, and will be treated with the corresponding dose. This study is designed to assess the preliminary efficacy and safety of MHB036C monotherapy in subjects with some types of advanced or metastatic solid tumors, so as to determine the recommended phase 2 dose (RP2D); and to assess the immunogenicity and pharmacokinetic profiles of MHB036C.

ELIGIBILITY:
Inclusion Criteria:

Participants enrolled must meet all of the following criteria:

General conditions

1. Participants voluntarily agree to participate in the study and sign the Informed Consent Form (ICF).
2. Participants aged 18 years or older (inclusive), without gender limitation.
3. Participants with ECOG performance score of 0 ~ 1.
4. Participants with expected survival time of more than 3 months.
5. Eligible participants of childbearing potential (males and females) must agree to take reliable contraceptive measures (hormone or barrier method, or absolute abstinence, etc.) with their partners during the study and within at least 90 days after the last dose; female participants of childbearing potential must have a negative results of blood pregnancy test within 7 days before the first dose of the investigational product, and must be non-lactating.
6. Participants who are able to understand study requirements, and willing and able to comply with arrangements of study and follow-up procedures.

   Neoplasm-related criteria
7. Participants to be enrolled in part one must have histologically or cytologically confirmed advanced or metastatic solid tumors, which have failed or are intolerant to standard of care (SOC), or for which no SOC is available;
8. Participants to be enrolled in part two must have histologically or cytologically confirmed advanced or metastatic solid tumors, including but not limited to the following types: non-small cell lung cancer (NSCLC); small cell lung cancer (SCLC); pancreatic ductal adenocarcinoma (PDAC); head and neck squamous cell carcinoma (HNSCC); esophageal squamous cell carcinoma (ESCC); urothelial carcinoma (UC); ovarian cancer (OC); endometrial cancer (EC); breast cancer (BC); gastric cancer (GC); castration-resistant prostate cancer (CRPC); sweat gland carcinoma (SGC).

   1. Additional criteria for enrollment of participants with NSCLC:

      * Participants with unresectable advanced NSCLC who have failed standard of care with platinum doublet chemotherapy and immune-checkpoint inhibitors (ICIs), and are not suitable for radical therapy (NSCLC participants with driver gene mutations should have failed or are intolerant to targeted therapy for the corresponding driver gene mutation, or unsuitable for the corresponding targeted therapy as per investigator's evaluation ).
   2. Additional criteria for enrollment of participants with SCLC:

      * Participants with unresectable or metastatic SCLC who have previously received at least one line of systemic chemotherapy, including platinum-based chemotherapy and immune-checkpoint inhibitors (ICIs)
   3. Additional criteria for enrollment of participants with PDAC:

      * Participants with unresectable or metastatic PDAC who have previously received at least one line of systemic chemotherapy, including any stage in neoadjuvant/adjuvant/ palliative therapy
   4. Additional criteria for enrollment of participants with HNSCC:

      * Participants with unresectable advanced or metastatic HNSCC who have previously received at least one line of systemic chemotherapy, including platinum-based chemotherapy and ICIs (combined or sequential therapy).
   5. Additional criteria for enrollment of participants with ESCC:

      * Participants with unresectable or metastatic ESCC who have previously received at least one line of systemic chemotherapy (platinum-based chemotherapy).
   6. Additional criteria for enrollment of participants with UC:

      * Participants with unresectable, locally progressed, or metastatic (histologically including transitional cells and mixed of transitional/non-transitional cells) UC (sites of occurrence including renal pelvis, ureter, bladder, and urethra) who have previously received at least one line of chemotherapy, including platinum-based chemotherapy and ICIs (combined or sequential therapy).
   7. Additional criteria for enrollment of participants with OC:

      * Participants with OC (including rare types of epithelial ovarian cancer stipulated in the NCCN guidelines as well as fallopian tube cancer and primary peritoneal cancer) who had tumor recurrence or metastasis after receiving at least one line of platinum-based chemotherapy
   8. Additional criteria for enrollment of participants with EC:

      * Participants with recurrent or incurable EC who had tumor recurrence or progression following previous radical therapy, and subsequently received therapies including standard systemic therapy.
   9. Additional criteria for enrollment of participants with BC:

      * For participants with advanced/unresectable or metastatic TNBC: Participants who have received at least 1 line of systemic chemotherapy with anthracyclines and taxanes included in the prior systemic therapy (regardless of neoadjuvant/adjuvant/palliative therapy).
      * For BC participants with hormone receptor (HR) positive (ER+ and/or PR+) and HER2 expression negative (IHC 0, 1+ or IHC 2+ with ISH-): Participants who are intolerant or resistant to endocrine therapy, or unsuitable for endocrine therapy as per investigator's evaluation.
      * For BC participants with HER2 expression positive (IHC 3+ or IHC 2+ with ISH+): Participants who have previously received at least 1 line of therapy, which included HER2-targeted therapy.
   10. Additional criteria for enrollment of participants with GC:

       * Participants with unresectable or metastatic GC who have previously received at least one line of standard systemic chemotherapy, while the previous treatment regimens of HER2-positive (IHC 3+ or IHC 2+ with ISH+) participants must include HER2-targeted therapy.
   11. Additional criteria for enrollment of participants with CRPC:

       * Absence of neuroendocrine differentiation or small cell histology confirmed by histopathology;
       * Underwent surgical or medical castration, with testosterone levels below 50 ng/dL;
       * Objective progression as determined by radiographic progression after androgen deprivation therapy;
       * Participants has relapsed or progressed after receiving at least one of the following medications: abiraterone, enzalutamide, apalutamide, or darolutamide;
       * Participants has relapsed or progressed after previously docetaxel-based or mitoxantrone-based cytotoxic chemotherapy for metastatic CRPC;
       * Participants with at least 1 documented lesion confirmed by either a bone scan or a CT/MRI scan.
   12. Sweat gland carcinoma (SGC): unresectable or metastatic SGC.
9. Participants who agree to provide the pre-treatment tumor tissue samples for retrospective testing of target expression and other biomarkers (participants who agree but are unable to provide pre-treatment tumor tissue sample may also be enrolled). Expression of target in tumor tissue samples collected from participants will not be used as a criterion for participant enrollment.
10. Participants with at least one measurable tumor lesion as per RECIST v1.1 (generally, tumor lesions located in a previously irradiated areas or other locoregional treatment sites will not be considered as measurable lesions, unless the lesions have clearly progressed or still persist three months after radiotherapy); for participants with CRPC, evaluable lesions as defined by PCWG3 criteria, or at least one measurable tumor lesion as per RECIST v1.1 are required.

    Adequate bone marrow reserve and organ functions:
11. Adequate bone marrow reserve (without transfusion, treatment of colony-stimulating factor, or biologics with similar effects within 7 days prior to the screening);

    * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
    * Platelet count ≥ 100 × 109/L;
    * Hemoglobin ≥ 9.0 g/dL.
12. Adequate hepatic function (with reference to normal values specified by the clinical study site):

    * Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); TBIL ≤ 2.0 × ULN if Gilbert's syndrome is present; TBIL ≤ 3.0 × ULN is permitted if direct bilirubin (DBIL) suggests extrahepatic obstruction.
    * For participants with non-hepatic tumors and without hepatic metastases, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) shall be ≤ 3.0 × ULN; for participants with hepatic tumors or hepatic metastases, AST and ALT shall be ≤ 5.0 × ULN;
13. Adequate renal function (with reference to normal values specified by the clinical study site):

    * Creatinine (Cr) ≤ 1.5 × ULN; when Cr > 1.5 × ULN, only participants with creatinine clearance (Ccr) ≥ 50 mL/min can be enrolled (using Cockcroft-Gault formula);
14. Adequate coagulation function:

    * Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, and international normalized ratio (INR) ≤ 1.5.
15. Adequate cardiac function:

    * Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram within 28 days prior to enrollment;
    * New York Heart Association (NYHA) Class < grade 3.

Exclusion Criteria:

Participants will be not enrolled if they meet any of the following exclusion criteria:

Neoplasm-related criteria:

1. Participants with 2 or more malignancies (except effectively treated non-melanoma skin cancer, cervical carcinoma in situ or other tumors, or malignancies considered cured) within 5 years prior to sign the Informed Consent Form.
2. Participants who have received chemotherapy within 3 weeks prior to the first dose of investigational product, or have received target therapy within 2 weeks prior to the first dose, or have received anti-tumor therapy including radiation therapy, biologic therapy, endocrine therapy, immunotherapy, etc. within 4 weeks prior to the first dose; or participants with the following conditions:

   * Medication of nitrosourea or mitomycin C within 6 weeks prior to the first dose of MHB036C;
   * Medication of oral fluoropyrimidines or small molecule targeted agents within 5 half-lives of such drug before first dose of investigational product.
   * Medication of traditional Chinese medicine with anti-tumor indications within 2 weeks prior to the first dose of investigational product.
3. Medication of other unmarketed investigational products or therapies within 4 weeks prior to the first dose of investigational product.
4. Presence of brain metastases and/or carcinomatous meningitis. Participants previously treated for brain metastases may be considered to be enrolled in this study, provided they have been in stable condition for at least 1 month, have no progression confirmed by radiographic examination within 4 weeks prior to the first dose of investigational product, all neurological symptoms have recovered, no evidence of new or enlarging brain metastases, and radiation or surgical had been discontinued for at least 14 days prior to the first dose of investigational product, or with steroid therapy ≤10 mg/day prednisone or equivalent dose of similar drugs within 14 days prior to the first dose of investigational product or during the study. This exception does not include carcinomatous meningitis, which should be excluded regardless of clinical stability.
5. Participants previously received same targeted therapy will be excluded.
6. Participants with adverse reactions from previous anti-tumor therapy that have not recovered to ≤Grade 1 as per CTCAE 5.0 (except for toxicities without safety risks as determined by the investigator, such as alopecia, hypothyroidism stably managed by hormone replacement therapy, etc.).

   General conditions:
7. Participants underwent major organ surgery (excluding biopsy) or significant trauma within 4 weeks prior to the first dose of investigational product or require elective surgery during the study.
8. Participants vaccinated with attenuated live vaccines (except for SARS-CoV-2 vaccination) within 4 weeks prior to the first dose of investigational product.
9. Participants received treatment with systemic corticosteroids (prednisone at > 10 mg/day, or similar drugs at equivalent dose) or other immunosuppressive agents within 14 days prior to the first dose of investigational product, with the following exceptions:

   * Treatment with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids;
   * Short-term use of glucocorticoids for prophylaxis (e.g., prevention of contrast media allergy).
10. Participants with clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder, or any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement, or prior pneumonectomy.
11. Participants with history of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, or has current ILD/pneumonitis, or where suspected ILD/pneumonitis that cannot be ruled out by imaging examination at screening.
12. Participants with active pulmonary tuberculosis.
13. Participants with clinically diagnosed corneal disease.
14. Participants with current active infection requiring systemic therapy.
15. Participants with positive results in virus serology tests (participants receiving antiviral prophylaxis other than interferon are allowed to be enrolled):

    * anti-HIV antibody positive;
    * Or, positive results of both HBsAg and HBV-DNA (i.e., HBV-DNA result is not below the LOD);
    * Or, positive results of both HCV Ab and HCV-RNA (i.e., HCV-RNA result is not below the LOD).
16. History of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    * Severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, or second-degree to third-degree atrioventricular block;
    * Fridericia-corrected QT interval (QTcF) > 450 ms for males or > 470 ms for females;
    * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke and other major cardiovascular and cerebrovascular events within 6 months prior to the first dose;
    * New myocardial infarction or unstable angina within 6 months prior to enrollment;
    * Clinically uncontrolled hypertension;
17. Participants with active autoimmune disorders (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for participants with clinically stable autoimmune thyroid disease or type I diabetes mellitus.
18. Participants with clinically uncontrolled effusion in third spacing, deemed as inappropriate for enrollment by the investigator.
19. Participants known to have hypersensitivity or delayed hypersensitivity to certain components or analogues of the study drug.
20. Participants with drug abuse or any other medical conditions, such as clinically significant cardiac or psychological conditions that, in the opinion of the investigator, may interfere with study participation or the results of the clinical study.
21. Participants known to have alcohol or drug abuse.
22. Females who are pregnant or lactating, or males/females who plan for childbirth.
23. Participants who are estimated to have poor compliance in study participation, or unsuitable to participate this clinical study by the opinion of the investigator for the history of other serious systemic disorders, or with other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-23 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | From the day of the first dose of MHB036C to 30 days after the day of the last dose of MHB036C
  Adverse events was assessed by investigator(s) according to NCI-CTCAE v5.0
Number of participants with dose-limiting toxicities | 21 days after the first dose of MHB036C
  Dose-limiting toxicities are defined as side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter: Maximum concentration (Cmax) | Within 5 cycles (each cycle is 21 days)
  Categories: MHB036C, total antibody, free toxin MH30010008
PK parameter: Time to maximum concentration (Tmax) | Within 5 cycles (each cycle is 21 days)
  Categories: MHB036C, total antibody, free toxin MH30010008
PK parameter: Area under the concentration-time curve (AUC) | Within 5 cycles (each cycle is 21 days)
  Categories: MHB036C, total antibody, free toxin MH30010008
PK parameter: Trough concentration (Ctrough) | Within 5 cycles (each cycle is 21 days)
  Categories: MHB036C, total antibody, free toxin MH30010008
PK parameter: Terminal or apparent terminal half-life (t1/2) | Within 5 cycles (each cycle is 21 days)
  Categories: MHB036C, total antibody, free toxin MH30010008
PK parameter: Systemic clearance (CL) | Within 5 cycles (each cycle is 21 days)
  Categories: MHB036C, total antibody, free toxin MH30010008
Immunogenicity Assessment | Within 5 cycles (each cycle is 21 days)
  Assessment of anti-drug antibody (ADA)
Objective Response Rate (ORR) | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Duration of Response (DOR) | 24 months
  DOR was defined as the time from first assessment of PR or CR until disease progression.
Disease Control Rate (DCR) | 24 months
  DCR was defined as the proportion of participants with a complete response (CR), partial response (PR) or stable disease (SD).
Progression Free Survival (PFS) | 24 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Pindara Private Hospital, Gold Coast, Queensland
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia
  - Cabrini Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided